CLINICAL TRIAL: NCT01683383
Title: A Randomized Clinical Trial of Therapeutic Hypothermia During Transport for Hypoxic Ischemic Encephalopathy (HIE): Device-regulated Cooling Versus Standard Practice.
Brief Title: California Transport Cooling Trial
Acronym: CTCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Inspiration Healthcare (Other)
Responsible Party: Principal Investigator, Krisa P Van Meurs, Professor of Pediatrics, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22993
Record Dates: First submitted 2012-09-06; First posted 2012-09-11 (Estimated); Results first posted 2014-12-08 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Hypoxic Ischemic Encephalopathy
Keywords: Hypoxic ischemic encephalopathy; Therapeutic hypothermia; Whole body cooling; Transport cooling
MeSH Terms: conditions — Hypoxia-Ischemia, Brain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (standard practice) (Active Comparator): Subjects in Arm 1 will receive passive or active cooling as per center practice with rectal temperatures being recorded every 15 minutes.
  Interventions: Other: Control (standard practice)
- Device (servo-regulated cooling) (Experimental): Subjects in Arm 2 will be placed on cooling blanket connected to the Tecotherm Neo (Inspiration Healthcare LTD UK). Temperature will be monitored continuously and servo-regulated using a rectal temperature probe.
  Interventions: Device: Device (servo-regulated cooling)

INTERVENTIONS:
Device: Device (servo-regulated cooling) — Subjects in Arm 2 will be placed on cooling blanket connected to the Tecotherm Neo (Inspiration Healthcare LTD UK). Temperature will be monitored continuously and servo-regulated using a rectal temperature probe.
  Other Names: Tecotherm Neo
  Arms: Device (servo-regulated cooling)
Other: Control (standard practice) — Subjects in Arm 1 will receive passive or active cooling as per center practice with rectal temperatures being recorded every 15 minutes.
  Arms: Control (standard practice)

SUMMARY:
Hypoxic ischemic encephalopathy (HIE) remains a major cause of death and severe disability despite advances in neonatal and perinatal medicine. Therapeutic hypothermia is the single most promising intervention for HIE. Reduction of brain temperature by 2° to 5°C has shown to be neuroprotective in newborn and adult animal models of brain ischemia. Therapeutic hypothermia instituted within 6 hours of birth has been shown to significantly improve survival and neurodevelopmental outcome in term newborns with HIE. Hypothermia is most effective if begun during the latent period, before the secondary energy failure. It is not known whether cooling initiated after 6 hours of age is effective.

The goal of this proposal is to test the efficacy of the cooling device in achieving the target temperatures in patients with moderate to severe HIE during transport when compared with current practices.

DETAILED DESCRIPTION:
Statement of the Problem:

Hypoxic ischemic encephalopathy (HIE) remains a major cause of death and severe disability despite advances in neonatal and perinatal medicine. Therapeutic hypothermia is the single most promising intervention for HIE. Reduction of brain temperature by 2° to 5°C has shown to be neuroprotective in newborn and adult animal models of brain ischemia. Therapeutic hypothermia instituted within 6 hours of birth has been shown to significantly improve survival and neurodevelopmental outcome in term newborns with HIE. Hypothermia is most effective if begun during the latent period, before secondary energy failure. It is not known whether cooling initiated after 6 hours of age is effective. Animal studies have shown that the sooner the initiation of cooling, the better the outcome. They have also suggested that the latent period may be shorter with a more severe insult. Cooling should be initiated as soon as possible, preferably within 2 hours and not later than 6 hours. There have been six large randomized clinical trials supporting the efficacy of therapeutic hypothermia for HIE and it is now the standard of care in the U.S. and internationally.

Once a patient qualifies for cooling, whole body cooling or selective head cooling is initiated. However, most birth hospitals do not have the ability to provide therapeutic hypothermia; thus, patients must be transported to Level 3 NICUs specially equipped to provide this therapy. As there is a limited therapeutic window for induction of hypothermia, it would be ideal to initiate therapeutic hypothermia as soon as the patient qualifies for cooling therapy. If cooling is initiated at the birth hospital, neuroprotective temperatures can be achieved several hours prior to arrival in the cooling center.

At this time patients cooled in transport receive passive cooling (turning off the active warming devices such as the transport isolette) or active cooling (ice packs placed around the baby). These practices have been shown to present a significant risk for over-cooling and under-cooling. The risks associated with excessive cooling include bradycardia, cardiac arrest, and coagulation disturbances. Undercooling likely results in reduced efficacy of the neuroprotective effects provided by therapeutic hypothermia.

Primary and secondary endpoints Primary end point: The percentage of temperatures in the target range (33°-34°C) both within and between enrolled infants after cooling initiation by the transport team.

Secondary end point: Time to the target temperature range (33°-34°C), percentage of newborns in target temperature range one hour after cooling initiation by transport team, and temperature ranges.

Study Design The proposed California Transport Cooling Trial (CTCT) is a prospective randomized multi-center clinical trial to be conducted by nine transport teams based at level III NICUs in California who perform therapeutic hypothermia for HIE. The on-call neonatologist at the participating cooling center will determine if the infant qualifies for cooling. Infants greater than or equal to 35 weeks and less than six hours of age who are being transported to a cooling center will be eligible. The transport team will randomize the infant to either cooling as per center practice (Arm 1) or device-regulated cooling (Arm 2). Subjects in Arm 1 will receive passive or active cooling as per center practice with rectal temperatures being recorded every 15 minutes. Subjects in Arm 2 will be placed on cooling blanket connected to the Tecotherm Neo. Temperature will be monitored continuously and servo-regulated using a rectal temperature probe. Pertinent clinical data will be collected using CPQCC/CPeTS data forms and CTCT data forms. Temperatures from initiation of cooling until admission to the cooling center will be analyzed for percentage of temperatures in the target range after cooling initiation by the transport team, time to target temperature range, percentage of newborns in the target temperature range 1 hour after cooling initiation by the transport team, and temperature ranges. ANOVA method will be used to compare the temperature ranges across arms. Cox proportional hazard model will be used to compare time to target temperature. Safety outcomes will be compared using standard logistic regression.

Study Methods Subjects assigned to Arm 1 will be cooled as per the usual center practice with recording of rectal temperatures every 15 minutes. Arm 2 subjects will be cooled using a portable servo-regulated cooling device using a rectal probe. Temperatures will be stored on the memory card every minute. No PHI will be stored in the cooling device. Data will be downloaded from the device at the conclusion of the transport.

Sample Size and Estimated Study Duration Power calculations for this study were based on anticipated 140 patients requiring initiation of therapeutic hypothermia by nine transport teams over a period of one year. A 70% consent rate and 50 patients per arm will provide 90% power to detect 30% absolute difference in the percentage of temperatures in the target range assuming a standard deviation for percentage of temperature in the target range of 45% based on the Kendall study, published in Archives of Diseases of Childhood in 2010. All analyses will adjust for center and will be two-sided and conducted at the 0.05 level of significance.

We estimate that patient enrollment will take approximately one year. Data analysis, manuscript preparation, and submission will be completed within 6 months of completion of enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Term or near-term infants with gestational age ≥35 weeks who meet institutional criteria for use of therapeutic hypothermia and in whom the decision has been made to perform cooling during transport.

Exclusion Criteria:

* Presence of a congenital or lethal chromosomal anomaly
* Decision to not provide full intensive care
* Refusal to consent

Max Age: 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2012-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Krisa Van Meurs, M.D., Principal Investigator — Stanford University
Locations (9):
- United States (9):
  - Loma Linda University Children's Hospital, Loma Linda, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital & Research Center, Oakland, California
  - Kaiser Permanente Oakland/Walnut Creek, Oakland, California
  - Stanford University, Palo Alto, California
  - Sutter Medical Center, Sacramento, California
  - Rady Childrens Hospital, San Diego, California
  - University of California San Francisco Medical Center, San Francisco, California
  - Santa Clara Valley Medical Center, San Jose, California

REFERENCES:
- [Background] Gunn AJ, Gunn TR, de Haan HH, Williams CE, Gluckman PD. Dramatic neuronal rescue with prolonged selective head cooling after ischemia in fetal lambs. J Clin Invest. 1997 Jan 15;99(2):248-56. doi: 10.1172/JCI119153. PMID 9005993
- [Background] Vannucci RC, Perlman JM. Interventions for perinatal hypoxic-ischemic encephalopathy. Pediatrics. 1997 Dec;100(6):1004-14. doi: 10.1542/peds.100.6.1004. No abstract available. PMID 9374573
- [Background] Gluckman PD, Williams CE. When and why do brain cells die? Dev Med Child Neurol. 1992 Nov;34(11):1010-4. doi: 10.1111/j.1469-8749.1992.tb11407.x. No abstract available. PMID 1358734
- [Background] Iwata O, Iwata S, Thornton JS, De Vita E, Bainbridge A, Herbert L, Scaravilli F, Peebles D, Wyatt JS, Cady EB, Robertson NJ. "Therapeutic time window" duration decreases with increasing severity of cerebral hypoxia-ischaemia under normothermia and delayed hypothermia in newborn piglets. Brain Res. 2007 Jun 18;1154:173-80. doi: 10.1016/j.brainres.2007.03.083. Epub 2007 Apr 1. PMID 17475224
- [Background] Gluckman PD, Wyatt JS, Azzopardi D, Ballard R, Edwards AD, Ferriero DM, Polin RA, Robertson CM, Thoresen M, Whitelaw A, Gunn AJ. Selective head cooling with mild systemic hypothermia after neonatal encephalopathy: multicentre randomised trial. Lancet. 2005 Feb 19-25;365(9460):663-70. doi: 10.1016/S0140-6736(05)17946-X. PMID 15721471
- [Background] Eicher DJ, Wagner CL, Katikaneni LP, Hulsey TC, Bass WT, Kaufman DA, Horgan MJ, Languani S, Bhatia JJ, Givelichian LM, Sankaran K, Yager JY. Moderate hypothermia in neonatal encephalopathy: efficacy outcomes. Pediatr Neurol. 2005 Jan;32(1):11-7. doi: 10.1016/j.pediatrneurol.2004.06.014. PMID 15607598
- [Background] Shankaran S, Laptook AR, Ehrenkranz RA, Tyson JE, McDonald SA, Donovan EF, Fanaroff AA, Poole WK, Wright LL, Higgins RD, Finer NN, Carlo WA, Duara S, Oh W, Cotten CM, Stevenson DK, Stoll BJ, Lemons JA, Guillet R, Jobe AH; National Institute of Child Health and Human Development Neonatal Research Network. Whole-body hypothermia for neonates with hypoxic-ischemic encephalopathy. N Engl J Med. 2005 Oct 13;353(15):1574-84. doi: 10.1056/NEJMcps050929. PMID 16221780
- [Background] Azzopardi DV, Strohm B, Edwards AD, Dyet L, Halliday HL, Juszczak E, Kapellou O, Levene M, Marlow N, Porter E, Thoresen M, Whitelaw A, Brocklehurst P; TOBY Study Group. Moderate hypothermia to treat perinatal asphyxial encephalopathy. N Engl J Med. 2009 Oct 1;361(14):1349-58. doi: 10.1056/NEJMoa0900854. PMID 19797281
- [Background] Simbruner G, Mittal RA, Rohlmann F, Muche R; neo.nEURO.network Trial Participants. Systemic hypothermia after neonatal encephalopathy: outcomes of neo.nEURO.network RCT. Pediatrics. 2010 Oct;126(4):e771-8. doi: 10.1542/peds.2009-2441. Epub 2010 Sep 20. PMID 20855387
- [Background] Jacobs SE, Morley CJ, Inder TE, Stewart MJ, Smith KR, McNamara PJ, Wright IM, Kirpalani HM, Darlow BA, Doyle LW; Infant Cooling Evaluation Collaboration. Whole-body hypothermia for term and near-term newborns with hypoxic-ischemic encephalopathy: a randomized controlled trial. Arch Pediatr Adolesc Med. 2011 Aug;165(8):692-700. doi: 10.1001/archpediatrics.2011.43. Epub 2011 Apr 4. PMID 21464374
- [Background] Fairchild K, Sokora D, Scott J, Zanelli S. Therapeutic hypothermia on neonatal transport: 4-year experience in a single NICU. J Perinatol. 2010 May;30(5):324-9. doi: 10.1038/jp.2009.168. Epub 2009 Oct 22. PMID 19847186
- [Background] Hallberg B, Olson L, Bartocci M, Edqvist I, Blennow M. Passive induction of hypothermia during transport of asphyxiated infants: a risk of excessive cooling. Acta Paediatr. 2009 Jun;98(6):942-6. doi: 10.1111/j.1651-2227.2009.01303.x. PMID 19484830
- [Background] Akula VP, Davis AS, Gould JB, Van Meurs K. Therapeutic hypothermia during neonatal transport: current practices in California. Am J Perinatol. 2012 May;29(5):319-26. doi: 10.1055/s-0031-1295661. Epub 2011 Dec 5. PMID 22143969
- [Background] Kendall GS, Kapetanakis A, Ratnavel N, Azzopardi D, Robertson NJ; Cooling on Retrieval Study Group. Passive cooling for initiation of therapeutic hypothermia in neonatal encephalopathy. Arch Dis Child Fetal Neonatal Ed. 2010 Nov;95(6):F408-12. doi: 10.1136/adc.2010.187211. Epub 2010 Sep 24. PMID 20870910
- [Background] Akula VP, Gould JB, Davis AS, Hackel A, Oehlert J, Van Meurs KP. Therapeutic hypothermia during neonatal transport: data from the California Perinatal Quality Care Collaborative (CPQCC) and California Perinatal Transport System (CPeTS) for 2010. J Perinatol. 2013 Mar;33(3):194-7. doi: 10.1038/jp.2012.144. Epub 2012 Dec 6. PMID 23223159
- [Derived] Akula VP, Joe P, Thusu K, Davis AS, Tamaresis JS, Kim S, Shimotake TK, Butler S, Honold J, Kuzniewicz M, DeSandre G, Bennett M, Gould J, Wallenstein MB, Van Meurs K. A randomized clinical trial of therapeutic hypothermia mode during transport for neonatal encephalopathy. J Pediatr. 2015 Apr;166(4):856-61.e1-2. doi: 10.1016/j.jpeds.2014.12.061. Epub 2015 Feb 12. PMID 25684087

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 131 infants were screened for eligibility at nine participating NICUs between October 1, 2012 and September 27th, 2013. Eligible infants had a gestational age of at least 35 weeks, met institutional criteria for use of therapeutic hypothermia, and a decision had been made to initiate cooling in transport.
Pre-assignment Details: Infants were excluded if they had a lethal congenital or chromosomal anomaly, the decision had been made to not provide full intensive care, or there was refusal of consent. Of 131 infants screened for eligibility, 30 were excluded, and 101 consented and were randomized.
Groups:
- Control (Standard Cooling): Infants were cooled as per the birth hospital practice either passively (turning the radiant warmer /incubator off) and/or actively (ice or gel packs).
- Device (Servo-regulated Cooling): Infants were placed on a servo-controlled cooling blanket after a rectal or esophageal probe was inserted. The temperature was servo-controlled using the Tecotherm Neo (Inspiration Medical LTD, Leicester, UK) (Appendix 1; online only) with the target temperature set to 33.5°C.
Period: Overall Study
Arm/Group | Control (Standard Cooling) | Device (Servo-regulated Cooling)
Started | 50 | 51
Transported and Treated | 49 | 51
Completed | 49 | 51
Not Completed | 1 | 0
Not completed — Infant was not transported | 1 | 0

BASELINE CHARACTERISTICS:
Population: Eligible newborns
Groups:
- Total: Total of all reporting groups
Arm/Group | Control (Standard Cooling) | Device (Servo-regulated Cooling) | Total
Number analyzed (Participants) | 49 | 51 | 100
Age, Customized [Mean (Standard Deviation); unit: Hours] — Chronological age at cooling initiation at birth hospital (hours)
  Hours
    Chron. age at cooling initiation at birth hospital | 26 (6) | 28 (6) | 27 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 22 | 47
  Male | 24 | 29 | 53
Birth weight [Mean (Standard Deviation); unit: Grams] | 3397 (627) | 3321 (523) | 3358 (610)
Gestational age [Mean (Standard Deviation); unit: Weeks] | 39.1 (1.7) | 39.1 (1.7) | 39.1 (1.7)
Apgar scores @ 1 minute [Number; unit: Participants] — Apgar scores ≤5 at either 5 or 10 minutes can be due to acute hypoxia ischemia in the intrapartum period and as such are often one of the eligibility criteria for therapeutic hypothermia to treat HIE.
  Participants
    Apgar @ 1 min ≤ 5 | 47 | 42 | 89
    Apgar @ 1 min > 5 | 2 | 9 | 11
Apgar scores @ 5 minutes [Number; unit: Participants] — Apgar scores ≤5 at either 5 or 10 minutes can be due to acute hypoxia ischemia in the intrapartum period and as such are often one of the eligibility criteria for therapeutic hypothermia to treat HIE.
  Participants
    Apgar @ 5 min ≤ 5 | 42 | 38 | 80
    Apgar @ 5 min > 5 | 7 | 13 | 20
Apgar scores @ 10 minutes [Number; unit: Participants] — Apgar scores ≤5 at either 5 or 10 minutes can be due to acute hypoxia ischemia in the intrapartum period and as such are often one of the eligibility criteria for therapeutic hypothermia to treat HIE.
  Participants
    Apgar @ 10 min ≤ 5 | 27 | 24 | 51
    Apgar @ 10 min > 5 | 22 | 27 | 49
Delivery room resuscitation: Oxygen [Number; unit: Participants]
  Oxygen | 46 | 47 | 93
  No oxygen | 3 | 4 | 7
Delivery room resuscitation: CPAP [Number; unit: Participants]
  CPAP | 18 | 16 | 34
  No CPAP | 31 | 35 | 66
Delivery room resuscitation: Bag and mask [Number; unit: Participants]
  Bag and mask | 43 | 43 | 86
  No bag and mask | 6 | 8 | 14
Delivery room resuscitation: Intubation with ventilation [Number; unit: Participants]
  Intubation with ventilation | 34 | 32 | 66
  No intubation with ventilation | 15 | 19 | 34
Delivery room resuscitation: Epinephrine [Number; unit: Participants]
  Epinephrine | 13 | 10 | 23
  No epinephrine | 36 | 41 | 77
Delivery room resuscitation: Chest compressions [Number; unit: Participants]
  Chest compressions | 20 | 22 | 42
  No chest compressions | 29 | 29 | 58
Respiratory support @ randomization: Non-invasive ventilation [Number; unit: Participants]
  Non-invasive ventilation: Yes | 15 | 9 | 24
  Non-invasive ventilation: No | 34 | 42 | 76
Respiratory support @ randomization: Conventional mechanical ventilation [Number; unit: Participants]
  Conventional mechanical ventilation: Yes | 26 | 29 | 55
  Conventional mechanical ventilation: No | 23 | 22 | 45
Respiratory support @ randomization: High-frequency ventilation [Number; unit: Participants]
  High-frequency ventilation: Yes | 3 | 4 | 7
  High-frequency ventilation: No | 46 | 47 | 93
Respiratory support @ randomization: Inhaled nitric oxide [Number; unit: Participants]
  Inhaled nitric oxide: Yes | 2 | 4 | 6
  Inhaled nitric oxide: No | 47 | 47 | 94
Pressors at randomization [Number; unit: Participants]
  Pressors used | 3 | 4 | 7
  No pressors used | 46 | 47 | 93
Cord gas: pH [Mean (Standard Deviation); unit: pH] | 6.91 (0.20) | 7.01 (0.15) | 6.96 (0.18)
Cord gas: base deficit [Mean (Standard Deviation); unit: mEq/L] | 15.6 (7.1) | 14.0 (4.7) | 14.8 (6.0)
First postnatal gas: pH [Mean (Standard Deviation); unit: pH] | 7.06 (0.20) | 7.02 (0.19) | 7.04 (0.19)
First postnatal gas: base deficit [Mean (Standard Deviation); unit: mEq/L] | 17.0 (6.7) | 17.5 (6.9) | 17.3 (6.8)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Temperatures in Target Range During Transport
Description: The percentage of temperatures in the target range (33°-34°C) during transport after cooling initiation by the transport team.
Time Frame: Participants will be followed for the duration of neonatal transport from the birth hospital to the cooling center, an expected average of 4 hours
Population: Total patients in each study arm
Measure: Median (Inter-Quartile Range); unit: Percentage of temperatures
Groups:
- Control (Standard Cooling): Subjects in Arm 1 will receive passive or active cooling as per center practice with rectal temperatures being recorded every 15 minutes.
Arm/Group | Control (Standard Cooling) | Device (Servo-regulated Cooling)
Number analyzed (Participants) | 49 | 51
Percentage of temperatures | 0 [0 to 52] | 73 [17 to 88]
Statistical Analysis 1: Comparison: Control (Standard Cooling) vs Device (Servo-regulated Cooling); Test type: Superiority or Other; p < 0.001, Adjusted Wald estimation

2. Secondary Outcome: Time to Target Temperature
Description: Time to the target temperature range (33°-34°C) from initiation of cooling by the transport team
Time Frame: as for outcome 1
Population: Total patients in each study arm
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Control (Standard Cooling) | Device (Servo-regulated Cooling)
Number analyzed (Participants) | 49 | 51
Minutes | 63 (37) | 44 (31)
Statistical Analysis 1: Comparison: Control (Standard Cooling) vs Device (Servo-regulated Cooling); Test type: Superiority or Other; p = 0.04, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Percentage of Participants in the Target Range at 1 Hour
Description: Percentage of participants in target range (33°-34°C) one hour after cooling initiation by the transport team
Time Frame: as for outcome 1
Population: Total participants in each study arm, excluding 8 participants in the control arm and 12 participants in the device arm who completed transport in < 1 hour.
Measure: Number; unit: Percentage of participants
Arm/Group | Control (Standard Cooling) | Device (Servo-regulated Cooling)
Number analyzed (Participants) | 41 | 39
Percentage of participants | 8 | 28

4. Secondary Outcome: Participants in Target Temperature Range Anytime During Transport
Description: Participants in target temperature range (33-34 C) anytime during transport
Time Frame: as for outcome 1
Population: Total participants in each study arm
Measure: Number; unit: Participants
Arm/Group | Control (Standard Cooling) | Device (Servo-regulated Cooling)
Number analyzed (Participants) | 49 | 51
Participants | 24 | 41
Statistical Analysis 1: Comparison: Control (Standard Cooling) vs Device (Servo-regulated Cooling); Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

5. Other Pre Specified Outcome: Safety Outcomes
Description: The incidence, intervention and outcome of cardiac arrhythmia, major bleeding, altered skin integrity, pulmonary hypertension, device-related events, death, and other serious adverse events from the time of initiation of transport cooling to the time of completion will be monitored.
Time Frame: as for outcome 1
Population: Total participants in each study arm
Measure: Number; unit: Participants
Arm/Group | Control (Standard Cooling) | Device (Servo-regulated Cooling)
Number analyzed (Participants) | 49 | 51
Participants
  Cardiac arrhythmia | 0 | 0
  Major bleeding (pulmonary hemorrhage) | 0 | 1
  Altered skin integrity | 0 | 0
  Pulmonary hypertension | 0 | 0
  Device-related events | 0 | 2
  Death | 6 | 9

ADVERSE EVENTS:
Time Frame: Data were collected from the time of initiation of cooling (Arm 1 or Arm 2) to admission at the cooling center
Arm/Group | Control (Standard Cooling) | Device (Servo-regulated Cooling)
Serious Adverse Events (participants affected / at risk) | 6/49 | 10/51
Other Adverse Events (participants affected / at risk) | 0/49 | 2/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (Standard Cooling) (N=49) | Device (Servo-regulated Cooling) (N=51)
Pulmonary hemorrhage (Vascular disorders) | 0 (0) | 1 (1) — Note: Pulmonary hemorrhage was present prior to randomization and was not attributable to the study intervention.
Death (General disorders) | 6 (6) | 9 (9) — Note: These deaths were all attributed to disease complications and were not attributable to the study intervention.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (Standard Cooling) (N=49) | Device (Servo-regulated Cooling) (N=51)
Equipment alarms (General disorders) | 0 (0) | 2 (2) — Brief equipment alarms when non-physiologic changes in temperature were registered by the device

LIMITATIONS AND CAVEATS:
1, The criteria used to initiate hypothermia varied. 2, Operational errors occurred in 9 newborns during device regulated cooling. 3, 9.6% of temperatures in the control arm were missing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No